CLINICAL TRIAL: NCT00002786
Title: PHASE I STUDY TO EVALUATE THE SAFETY OF CELLULAR ADOPTIVE IMMUNOTHERAPY USING GENETICALLY MODIFIED AND UNMODIFIED AUTOLOGOUS CD8+ TYROSINASE-SPECIFIC T CELLS FOR PATIENTS WITH METASTATIC MELANOMA
Brief Title: Biological Therapy in Treating Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 1017.01; FHCRC-1017.01; NCI-V96-0920; CDR0000064846 (Registry Identifier: PDQ); NCT00029419 (obsolete NCT alias)
Record Dates: First submitted 1999-11-01; First posted 2003-05-26 (Estimated); Last update posted 2010-05-10 (Estimated); Status verified 2010-05

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — aldesleukin

INTERVENTIONS:
Biological: aldesleukin
Biological: therapeutic tumor infiltrating lymphocytes

SUMMARY:
RATIONALE: Biological therapies use different ways to stimulate the immune system and stop cancer cells from growing.

PURPOSE: Phase I/II trial to study the effectiveness of biological therapy in treating patients who have metastatic melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the safety and toxicity of cellular adoptive immunotherapy using autologous CD8+ antigen-specific T-cell clones in patients with metastatic melanoma.
* Estimate the duration of in vivo persistence of adoptively transferred CD8+ antigen-specific cytotoxic T-cell clones in these patients.
* Evaluate the antitumor effects of CD8+ antigen-specific T-cell clones in these patients.

OUTLINE: Autologous peripheral blood mononuclear cells are harvested and then CD8+ cytotoxic T-lymphocyte (CTL) clones targeting melanosomal antigens are generated ex vivo. Patients receive cellular adoptive immunotherapy comprising autologous CD8+ CTL clones over 30 minutes on day 1. Patients also receive interleukin-2 subcutaneously every 12 hours on days 1-14 of courses 2-3. Treatment repeats every 3 weeks for 3 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed for approximately 1 year after the last infusion.

PROJECTED ACCRUAL: Approximately 20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histopathologically proven metastatic melanoma

  * No CNS metastases
* HLA-A2 positive
* Bidimensionally measurable disease by palpation on clinical exam or radiographic imaging (x-ray, CT scan, or MRI)
* Surgically accessible site for tumor cell procurement (skin, subcutaneous nodule, or superficial node) and patient clinically eligible for such surgery

PATIENT CHARACTERISTICS:

Age

* 18 to 75

Performance status

* Karnofsky 80-100%

Life expectancy

* More than 16 weeks

Hematopoietic

* WBC greater than 4,000/mm^3
* Absolute neutrophil count greater than 2,000/mm^3
* Platelet count greater than 100,000/mm^3
* Hematocrit greater than 30%

Hepatic

* Bilirubin no greater than 1.6 mg/dL
* SGOT no greater than 150 IU (or no greater than 3 times normal)
* Prothrombin time no greater than 1.5 times control

Renal

* Creatinine no greater than 2.0 mg/dL
* Calcium no greater than 12 mg/dL

Cardiovascular

* No congestive heart failure
* No clinically significant hypotension
* No symptoms of coronary artery disease
* No arrhythmia on EKG requiring drug therapy

Pulmonary

* No severe chronic obstructive pulmonary disease
* FEV_1 at least 1.0 L
* DLCO at least 45% of predicted

Other

* No active infection or oral temperature greater than 38.2 degrees C within 72 hours of study
* No systemic infection requiring chronic maintenance or suppressive therapy
* HIV negative
* No history of seizures
* No retinitis or choroiditis
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use adequate contraception
* Peripheral blood samples available weekly for 4 consecutive weeks

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 4 weeks since other prior immunotherapy

Chemotherapy

* 1 or 2 courses of cytoreductive chemotherapy allowed for bulky disease
* At least 4 weeks since prior standard or investigational chemotherapy

Endocrine therapy

* At least 4 weeks since prior steroid therapy

Radiotherapy

* At least 4 weeks since prior radiotherapy

Surgery

* Not specified

Other

* At least 4 weeks since other prior investigational drug therapy and recovered

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 1995-10; Study Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cassian Yee, MD, Study Chair — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States